CLINICAL TRIAL: NCT02535390
Title: Action-Based Cognitive Remediation to Improve Vocational Outcomes in Depression
Acronym: ABCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Dr., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSYC-152-14
Record Dates: First submitted 2015-04-20; First posted 2015-08-28 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: cognitive remediation; vocational outcomes
MeSH Terms: conditions — Depression | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Action based cognitive remediation (Experimental): Participants in this condition will engage in simulated real world tasks in addition to standard cognitive remediation and group therapy sessions.
  Interventions: Behavioral: Action based cognitive remediation
- Standard cognitive remediation (Active Comparator): Participants in this condition will engage in computerized cognitive training exercises in addition to standard cognitive remediation and group therapy sessions.
  Interventions: Behavioral: Cognitive remediation

INTERVENTIONS:
Behavioral: Action based cognitive remediation — This is a novel form of cognitive remediation in which participants engage in simulated real world tasks in groups and receive therapist feedback in addition to receiving standard cognitive remediation.
  Arms: Action based cognitive remediation
Behavioral: Cognitive remediation — Cognitive remediation engages participants in computerized exercises meant to improve cognitive functions and provides therapist feedback for how these improvements manifest in everyday life.
  Arms: Standard cognitive remediation

SUMMARY:
Major depressive disorder places a tremendous burden on workplace disability each year. Its diagnosis is based on the presence of characteristic symptoms that include disturbances in mood regulation, maladaptive beliefs, and behaviour. Impairment in neurocognitive functions (e.g., information processing speed, attention, memory, problem solving skills) is absent from current diagnostic criteria and off the radar in most clinical treatment settings, yet increasingly recognized as a primary cause of poor work functioning and outcomes. This disconnect between the root causes of poor vocational outcomes and targets of treatment has resulted in a failure to return to work following illness, job underproductivity, and work-related stress, which contribute to indirect costs to society each year. The investigators seek to expand scientific support for treating neurocognitive impairments in order to increase occupational productivity and reduce job-related stress associated with depression. The investigators developed a novel group cognitive remediation (CR) treatment, Action-Based Cognitive Remediation (ABCR). It builds on procedural learning skills with explicit work-related role-plays to facilitate immediate and salient abstraction of drill and practice remediation techniques. The activities were developed in collaboration with a community rehabilitation partner in this study through systematic interviews with job placement specialists and supervisors from employment sites used by the agency. The props match those used in work settings and include miniature versions of a cash register, filing system, conveyer belt, cleaning closet, garden nursery, and secretarial station. The activities capitalize on procedural learning skills through roleplays and props that simulate a work environment. ABCR maintains important aspects of drill and practice, strategic monitoring to enhance flexible problem solving approaches, and bridging. The role-plays follow computerized drill and practice exercise and therapists facilitate group discussions of how cognitive skills and flexibility in thinking from drill and practice can be effective while directly engaged in an everyday work environment. Thus, bridging used in ABCR is a tangible, procedural, and realistic. This approach to bridging differentiates the treatment from standard CR, where the discussion-based approach is limited by the auditory learning, memory, and abstraction deficits observed in depression.

DETAILED DESCRIPTION:
Participants will meet with the PI or clinical graduate student to discuss components of cognitive remediation, expectations, and client goals. Follow-up meetings will occur to ensure client satisfaction and determine progress on goal achievement.

Randomization to ABCR or standard CR will be done in groups of 8 to ensure an adequate number of participants in each group. Twenty-four participants will be randomized to each group over the course of the study. Several aspects of the treatments are matched for ideal comparison. Both groups will meet two times per week, two hours per session, for 8 weeks. The same computerized drill and practice, strategic monitoring, and verbal bridging approaches will be used in both groups. The primary differences are the ratio of each aspect of treatment and the manner in which they are bridged work environment. In the standard CR group 60% of the sessions involve computerized drill and practice. In the ABCR group, only 20% of the group sessions are devoted to computer drills, whereas 40% involve the simulated work skills that are directly linked to those computer tasks (see Figure 1 for an example). The remaining 40% of both of the groups involve a didactic component that introduces concepts for that session (e.g., memory strategies, how to avoid distractors), review of homework, and group discussion of bridging. Strategic monitoring occurs during all aspects of treatment, though in ABCR the link between computerized drills and work is made explicit by moving back and forth from computer drills to the role-play tasks. Graduate students in a clinical psychology program who are trained and supervised by Dr. Bowie will conduct the treatment groups. These students will be blind to study hypotheses, though it will not be possible to blind them to the group. Video recordings of sessions are regularly reviewed with Dr. Bowie to ensure treatment fidelity.

In both groups, participants are given the opportunity to engage in supplemental homework exercises outside of the scheduled treatment groups. Scientific Brain Training Pro will be used for computer drills in session and for homework, a program the investigators have used in previous studies. The company provides its software for this research at no cost, but has no input into the design or output of this study. Due to the online availability of the exercises, participants are encouraged to login to the program one or two times per day for 20 minutes each session. Variability in homework completion is expected (and therefore considering it as a treatment process variable and potential mediator of longer-term durability and generalization), yet compliance with the sample is anticipated because they will be engaged standard vocational services programs four days per week, giving them access to an on-site computer room before or after attending their regular appointments.

Few previous studies have examined work stress as a function of supplemental treatments in vocational rehabilitation and to the investigators' knowledge this project will be the first to measure both self-reported and psychophysiological indicators of stress.

ELIGIBILITY:
Inclusion Criteria:

* DSM Axis 1 Mental disorder of Major Depressive Disorder
* Between the ages of 18 and 65 years old

Exclusion Criteria:

* Reading level below grade 6 (assessed with the Wide Range Achievement - Reading Recognition Test)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-12; Primary Completion 2018-06-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in composite scores on neurocognitive assessments | Assessed at baseline, immediately after treatment, and 1 year later
  Assessed with a standardized battery of tests sensitive to cognitive changes. Includes tests measuring domains of attention/vigilance, processing speed, working memory, verbal learning, visual learning, reasoning, and problem solving.

SECONDARY OUTCOMES:
Change in functional competence | Assessed at baseline, immediately after treatment, and 1 year later
  Assessed with the UCSD Performance-based Skills Assessment.
Change in work status | Assessed at baseline, immediately after treatment, and 1 year later
  Categorical analysis of work/role function: unemployed, part-time, full-time
Change in everyday real world functioning | Assessed at baseline, immediately after treatment, and 1 year later
  Assessed with the WHO-DAS

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowie, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada